CLINICAL TRIAL: NCT03347487
Title: Deep Brain Stimulation of the Bilateral Habenula for Treatment- Resistant Major Depression: An Open Label Pilot Trial
Brief Title: DBS of the Habenula for Treatment- Resistant Major Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 7 patients were included in this study which aimed for 13 participants. Preliminary data were sufficient for developing further study.
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Bomin Sun, Director of the Department of Functional Neurosurgery, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018 DBS-Hb MDD
Record Dates: First submitted 2017-11-11; First posted 2017-11-20 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Treatment Resistant Major Depression Disorder
Keywords: Bilateral Habenula; Treatment Resistant Major Depressive Disorder

STUDY DESIGN:
Intervention Model Description: All subjects will receive bilateral surgical implantation of DBS system.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deep Brain Stimulation of Bilateral Habenula (Experimental)
  Interventions: Procedure: Deep brain stimuation system implantation

INTERVENTIONS:
Procedure: Deep brain stimuation system implantation — All subjects will receive bilateral surgical implantation of DBS system.The Medtronic DBS 3389 electrode is utilized in this study. The DBS system includes a dual-channel neurostimulator kit, lead kit, extension kit, clinician-operated wireless programmer, test stimulator, and patient controller.
  Other Names: DBS; Activa RC System

SUMMARY:
The habenula(Hb) is an epithalamic structure located at the center of the dorsal diencephalic conduction system, a pathway involved in linking forebrain to midbrain regions. An increasing number of studies indicates that overactivity in the lateral habeluna(LHb) is present during depressed states, where it could drive the changes in midbrain activity linked to depression. Deep brain stimulation(DBS) of the major afferent bundle (i.e., stria medullaris thalami) of the LHb can treat treatment-resistant major depression(TRD). There is no clinical case of directly stimulating habeluna for treatment TRD. This research will investigate effectiveness and safety of bilateral DBS to habenula for patients with TRD. This study will also use structural and functional MRI to explore the underlying mechanism of Hb's effects on TRD.

ELIGIBILITY:
Inclusion Criteria:

* Men and women(non-pregnant) aged 18-65 years old;
* DSM-5 diagnosis (assessed by Structured Clinical Interview for DSM-5) of a current major depressive episode(MDE), either nonpsychotic unipolar major depressive disorder (MDD) or bipolar disorder (BD);
* Chronic illness with current MDE ≥ 24 months duration and/or recurrent illness with at least a total of 4 lifetime episodes (including current episode ≥ 12 months) and a minimum of 5 y since the onset of the first depressive episode;
* For subjects with a bipolar disorder: the last manic or hypomanic episode must have been ≥ 24 months before study enrollment and patients must be maintained on a mood stabilizer (e.g. lithium or another mood stabilizer approved for bipolar disorder)
* Treatment resistance defined as Failure of at least 3 adequate treatments from at least two distinctly different classes (SSRI, SNRI, NaSSA, TCA+, lithium-addition) for a period of 6-8 weeks. If diagnosed as bipolar, failure to respond to (or inability to tolerate) a minimum of three treatments approved for bipolar disorder, including lithium and at least one medication FDA-approved for bipolar depression (e.g., olanzapine/fluoxetine combination, quetiapine, lurasidone).
* At least 1 session of ECT, for which the series of ECT was terminated either due to adverse effects or insufficient response (including at least 6 sessions of bilateral ECT). Or unable to recieve ECT.
* Symptom Severity: HAMD-17 total ≥21;
* Stable antidepressant medical regimen for the month preceding surgery;
* Anticipates a stable psychotropic medication regimen in the next 12 months;
* Able and willing to give written informed consent;
* Modified mini-mental state examination (MMSE) score ≥ 27；

Exclusion Criteria:

* Schizophrenia /history of psychosis unrelated to MDD;
* Severe personality disorder (assessed by SCID-II);
* Alcohol or substance abuse/dependence within 6 months, excluding nicotine dependence;
* Current substantial suicidal risk as defined by a plan or clear immediate intent for self-harm, or had a serious suicide attempt within the last year;
* Neurological disease (e.g., Parkinson's disease)
* Any history of seizure disorder or hemorrhagic stroke;
* Abnormal brain MRI ;
* Previous sterosurgery;
* Any medical contraindication to surgery;
* Does not have adequate family/friend support as determined by psychological screening and/or interview;
* Unable to maintain a stable psychotropic medication regimen in the next 12 months;
* Pregnant or has plans to become pregnant in the next 12 months;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
changes in the Hamilton Depression Scale(HAMD-17) score from baseline to 9 months | Baseline (preoperative),one month, 3 months, 6 months, 9 months
  The score of the scale ranges from 0 to 50.
changes in the Montgomery-Asberg Depression Rating Scale from baseline to 9 months | Baseline (preoperative),one month, 3 months, 6 months, 9 months
  The score of the scale ranges from 0 to 60.

SECONDARY OUTCOMES:
changes in the brain activity | Baseline (preoperative),one month, 9 months
Side Effects | Baseline (preoperative),one month, 3 months, 6 months, 9 months
Young Mania Rating Scale (YMRS) | Baseline (preoperative),one month, 3 months, 6 months, 9 months
  YMRS is an eleven-item multiple choice diagnostic questionnaire which psychiatrists use to measure the severity of manic episodes. The score of the scale ranges from 0 to 60. Higher score means more severity of mania.
Changes in Hamilton Anxiety Scales(HAMA) | Baseline (preoperative),one month, 3 months, 6 months, 9 months
  Clinician administered assessment.The score of the scale ranges from 0 to 56.
Global Assessment of Functioning Scale(GAF) | Baseline (preoperative),one month, 3 months, 6 months, 9 months
  Clinician administered assessment.The score of the scale Scores range from 100 (extremely high functioning) to 1 (severely impaired).
Columbia Suicide Severity Rating Scale (C-SSRS) | Baseline (preoperative),one month, 3 months, 6 months, 9 months
  Clinician administered assessment.The Screener contains 6 "yes" or "no" questions in which respondents are asked to indicate whether they have experienced several thoughts or feelings relating to suicide over the past month and behaviors over their lifetime and past 3 months. Each question addresses a different component of the respondent's suicide ideation severity and behavior.
Changes in Beck Depression Inventory | Baseline (preoperative),one month, 3 months, 6 months, 9 months
  Self-rating scale. The score of the scale ranges from 0 to 63. Higher score means more severity of depression.
Chang in Pittsburgh Sleep Quality Index | Baseline (preoperative),one month, 3 months, 6 months, 9 months
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score ranging from 0 to 21. The high score means poor quality of sleep.
World Health Organization Quality of Life-BREF(WHO-BREF) | Baseline (preoperative),one month, 3 months, 6 months, 9 months
  The World Health Organization Quality of Life - BREF (WHOQOL-BREF) is a self-report questionnaire which assesses 4 domains of quality of life (QOL): physical health, psychological health, social relationships, and environment. It contains 26 items which is a 5 points scale. The higher score means better quality of life.
the MOS item short from health survey (SF-36) | Baseline (preoperative),one month, 3 months, 6 months, 9 months
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and are now widely utilized by managed care organizations and by Medicare for routine monitoring and assessment of care outcomes in adult patients. The higher score means better quality of life.
Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form | Baseline (preoperative),one month, 3 months, 6 months, 9 months
  The scoring of the Q-LES-Q-SF involves summing only the first 14 items to yield a raw total score. The last two items are not included in the total score but are stand-alone items. The raw total score ranges from 14 to 70.
Sheehan Disability Scale | Baseline (preoperative),one month, 3 months, 6 months, 9 months
  Self-rating scale. The SDS is a composite of three self-rated items designed to measure the extent to which three major domains in the patient's life are functionally impaired by psychiatric or medical symptoms. The SDS assesses functional impairment in three major life domains: work, social life/leisure activities, and family life/home responsibilities. The higher scores mean more severity of disability.
Changes in Neuropsychological measures(Scores of CANTAB tasks) | Baseline (preoperative),3 months, 9 months
  Neuropsychological measures contains six tasks which are Stop Signal Task, Spatial Working Memory, Paired Associated Learning, Stocking of Cambridge, Intra Extra dimensional Set Shifting, Reaction time Task

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ruijin Hospital Functional Neurosurgery, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Sartorius A, Kiening KL, Kirsch P, von Gall CC, Haberkorn U, Unterberg AW, Henn FA, Meyer-Lindenberg A. Remission of major depression under deep brain stimulation of the lateral habenula in a therapy-refractory patient. Biol Psychiatry. 2010 Jan 15;67(2):e9-e11. doi: 10.1016/j.biopsych.2009.08.027. No abstract available. PMID 19846068
- [Background] Sartorius A, Henn FA. Deep brain stimulation of the lateral habenula in treatment resistant major depression. Med Hypotheses. 2007;69(6):1305-8. doi: 10.1016/j.mehy.2007.03.021. Epub 2007 May 10. PMID 17498883
- [Background] Kiening K, Sartorius A. A new translational target for deep brain stimulation to treat depression. EMBO Mol Med. 2013 Aug;5(8):1151-3. doi: 10.1002/emmm.201302947. Epub 2013 Jul 4. No abstract available. PMID 23828711
- [Background] Dougherty DD, Rezai AR, Carpenter LL, Howland RH, Bhati MT, O'Reardon JP, Eskandar EN, Baltuch GH, Machado AD, Kondziolka D, Cusin C, Evans KC, Price LH, Jacobs K, Pandya M, Denko T, Tyrka AR, Brelje T, Deckersbach T, Kubu C, Malone DA Jr. A Randomized Sham-Controlled Trial of Deep Brain Stimulation of the Ventral Capsule/Ventral Striatum for Chronic Treatment-Resistant Depression. Biol Psychiatry. 2015 Aug 15;78(4):240-8. doi: 10.1016/j.biopsych.2014.11.023. Epub 2014 Dec 13. PMID 25726497
- [Background] Bergfeld IO, Mantione M, Hoogendoorn ML, Ruhe HG, Notten P, van Laarhoven J, Visser I, Figee M, de Kwaasteniet BP, Horst F, Schene AH, van den Munckhof P, Beute G, Schuurman R, Denys D. Deep Brain Stimulation of the Ventral Anterior Limb of the Internal Capsule for Treatment-Resistant Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2016 May 1;73(5):456-64. doi: 10.1001/jamapsychiatry.2016.0152. PMID 27049915
- [Derived] Huang Y, Sun B, Debarros J, Zhang C, Zhan S, Li D, Zhang C, Wang T, Huang P, Lai Y, Brown P, Cao C, Tan H. Increased theta/alpha synchrony in the habenula-prefrontal network with negative emotional stimuli in human patients. Elife. 2021 Jul 12;10:e65444. doi: 10.7554/eLife.65444. PMID 34251338